CLINICAL TRIAL: NCT04783467
Title: Feasibility and Acceptability of Time Restricted Eating (TRE) Among Endometrial Cancer Patients: the TREND Study
Brief Title: Time Restricted Eating (TRE) Among Endometrial Cancer Patients
Acronym: TREND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Mary Playdon, Assistant Professor, Investigator, University of Utah
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00126714
Record Dates: First submitted 2021-02-18; First posted 2021-03-05 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Trehalase; Appointments and Schedules

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating (TRE) Schedule (Experimental): For 6-weeks out of the 16-week randomized dietary crossover study, women will receive prepared frozen lunch and dinner meals as per the control schedule, but will be asked to consume daily meals, snacks, and calorie-containing beverages within an 8 to 10-hour period that fits their schedule. The meal plans will be individualized to meet weight maintenance energy requirements.
  Interventions: Behavioral: Time Restricted Eating (TRE) Schedule
- Control Schedule (No Intervention): For 4 weeks out of the 16-week randomized dietary crossover study, women will receive frozen lunch and dinner meals, and a standardized breakfast and snacks menu. The meal plans will be individualized to meet weight maintenance energy requirements. There are no restrictions on timing of eating.

INTERVENTIONS:
Behavioral: Time Restricted Eating (TRE) Schedule — [See arm/group descriptions]
  Arms: Time Restricted Eating (TRE) Schedule

SUMMARY:
The long-term goal of this study is to determine the efficacy of Time Restricted Eating (TRE) for improving metabolic health, preventing cardiometabolic comorbidities, and improving prognosis after endometrial cancer diagnosis. The primary objective of the protocol is to conduct a 16-week randomized dietary crossover study to evaluate the feasibility, fidelity and preliminary acceptability of TRE among endometrial cancer patients, and to provide proof of principle that TRE can improve metabolic health in this population.

DETAILED DESCRIPTION:
Enrollment: The study team will aim to recruit 15 endometrial cancer patients seen at the Huntsman Cancer Hospital Clinics. Consent may be completed via phone/email or in-person with the study clinical coordinator.

Dietary Intervention: Participants who are consented into the study will participate in a 16-week randomized dietary crossover intervention. The dietary intervention includes 5 study visits, and features a baseline visit, 2-week run-in period, 4-week control diet schedule with prepared frozen meals provided to participants, 4-week washout period, and a 6-week, 8 to 10-hour Time Restricted Eating (TRE) protocol (meal provision with 8 to 10-hour eating and 14 to 16-hour fasting periods). Women will be randomized to either control or TRE, then crossover to the other condition. For the control schedule, women will receive frozen lunch and dinner meals and be provided with a standardized breakfast and snacks menu, and there are no restrictions on timing of eating. For the TRE schedule, women will receive prepared frozen lunch and dinner meals as per the control schedule, but will be asked to consume daily meals, snacks, and calorie-containing beverages within an 8 to 10-hour period that fits their schedule. Fasting period will ramp up during the first week (e.g., Days 1-3, 12-14 h per day, Days 4-6, 14-16 h per day, Days 7+, 16 h per day). Women will be asked to schedule the eating period at the same time each day.

Study Visits and Assessments: Women will attend in-person study visits at the Huntsman Cancer Institute Center for Health Outcomes and Population Equity (HOPE).

* Baseline Visit (Visit 1): The clinical coordinator will obtain consent from the participant. Once consented, women will complete questionnaires to capture information on clinical and demographic factors, and chronotype. Height will be measured using stadiometer, weight will be measured using calibrated scales, waist circumference with measuring tape and blood pressure (BP) using an electronic BP monitor. Participants may take home questionnaires, with mailer, to complete at home.
* 2-Week Run-In Period: The purpose of the run-in period is to record women's usual times of eating episodes and appetite while following their habitual diet. Appetite will be measured using the MyCircacianClock (mCC) phone app that has the capability to sample subjects' current behaviors and experiences in real time in their natural environment. Women will complete 3 x 24-hour dietary recalls on non-consecutive days (ASA-24) and a physical activity recall (ACT24 available online or phone app, or via telephone conference with the clinical coordinator). Sleep and activity will also be objectively measured for 7-days using an Actiwatch.
* Visit 2: Women will provide fasting blood and stool samples. Weight, waist circumference and blood pressure will be measured.
* Control OR TRE Schedules: The participants will be expected to follow their randomized schedule for meal timing. During these schedules, for both study groups, participants will record timing of eating episodes daily using the MyCircadianClock app, complete 3 x 24-hour recalls (ASA24), 1 x ACT24 activity recall, and 7-days of sleep/physical activity will be objectively measured via Actiwatch.
* Visit 3: Women will provide fasting blood and stool samples. Weight, waist circumference and blood pressure will be measured.
* 4-Week Washout Period: During the washout period, women can return to their usual lifestyle. Meals will not be provided during this time.
* Visit 4: Visit 4 will include a telephone call only to discuss the next study phase and schedule meal provision.
* Visit 5: Women will provide fasting blood and stool samples. Weight, waist circumference and blood pressure will be measured. An exit interview may occur in person or via phone/video conference to ask questions about how well the intervention was tolerated and allow participants to provide feedback.
* Follow-Up: Approximately 6-months after consent and roughly 10 weeks after the end of the dietary intervention, participants will be asked to complete a follow-up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years or older
* Diagnosed with endometrial cancer (any stage)
* Clinically overweight or obese (BMI >= 25 kg/m2)
* At least 3 months post-cancer surgery and/or treatment
* Weight stable for 3 months prior to beginning the study (<4kg weight loss/gain)
* Have a cell phone that is able to download a phone App and able to use phone during the day

Exclusion Criteria:

* Persons with special dietary requirements
* Unable to provide informed consent
* Unable to read, write, or fill in questionnaires in English
* Insulin dependent diabetes
* Night shift workers
* Persons not able to use cell phone during day (like for work)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2021-10-07 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Women Referred that are Consented | From baseline to Visit 5 (Week 16)
  Feasibility of the TRE intervention will be measured be calculating the proportion (%) of women who were referred that were consented into the study. The study will be considered feasible of > 70% of participants are consented and retained.
Attrition as a Function of Time | From baseline to Visit 5 (Week 16)
  Number of participants who withdraw throughout the course of the study.
Percent of Scheduled Assessments Completed | From baseline to Visit 5 (Week 16)
  Feasibility of the TRE intervention will be assessed by calculating a percentage of scheduled biospecimen collection and questionnaires completed.
Number of TRE-Adherent Days per Week | From baseline to Visit 5 (Week 16)
  Feasibility of the TRE intervention will be measured by calculating the number of TRE-adherent days per week. Participants will be considered adherent if they fasted between 14-16 hours per day during the TRE phase according to the MCC App mealtime log. The study will be considered feasible if women adhere to the TRE protocol on average 5 days per week.
Fidelity of Time Restricted Eating (TRE) Intervention | From baseline to Visit 5 (Week 16)
  Fidelity will be evaluated as a percentage of protocol checklist items delivered as intended with a goal of 90%

SECONDARY OUTCOMES:
Change in blood pressure assessed via electronic blood pressure monitor | Baseline (Visit 1), Visit 2 (Week 2), Visit 3 (Week 6 or Week 8), Visit 5 (Week 16)
  Blood pressure will be taken using an electronic blood pressure monitor.
Change in waist circumference assessed via measuring tape | Baseline (Visit 1), Visit 2 (Week 2), Visit 3 (Week 6 or Week 8), Visit 5 (Week 16)
  Waist circumference will be measured using a measuring tape.
Change in BMI assessed via height and weight | Baseline (Visit 1), Visit 2 (Week 2), Visit 3 (Week 6 or Week 8), Visit 5 (Week 16)
  Participants' height and weight will be measured with stadiometer and electronic scales and used to calculate BMI.
Change in fasting blood glucose assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6 or Week 8), Visit 5 (Week 16)
  A small sample of blood will be taken from participants at designated study visits.
Change in HOMA-IR assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6 or Week 8), Visit 5 (Week 16)
  A small sample of blood will be taken from participants at designated study visits.
Change in c-peptide assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6 or Week 8), Visit 5 (Week 16)
  A small sample of blood will be taken from participants at designated study visits
Change in triglycerides assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6 or Week 8), Visit 5 (Week 16)
  A small sample of blood will be taken from participants at designated study visits
Change in HDL-cholesterol assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6 or Week 8), Visit 5 (Week 16)
  A small sample of blood will be taken from participants at designated study visits
Change in high sensitivity C-reactive protein assessed via blood draw | Visit 2 (Week 2), Visit 3 (Week 6 or Week 8), Visit 5 (Week 16)
  A small sample of blood will be taken from participants at designated study visits

CONTACTS AND LOCATIONS:
Overall Officials: Mary Playdon, PhD, MPH, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Agnew H, Kitson S, Crosbie EJ. Interventions for weight reduction in obesity to improve survival in women with endometrial cancer. Cochrane Database Syst Rev. 2023 Mar 27;3(3):CD012513. doi: 10.1002/14651858.CD012513.pub3. PMID 36971688